CLINICAL TRIAL: NCT04723212
Title: The Effect of Cognition and Age on Robotic Assessment of Upper Limb Passive and Active Sensory Processing
Brief Title: Robotic Assessment of Upper Limb Passive and Active Sensory Processing in Healthy Adults
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Geert Verheyden, Prof. Dr., KU Leuven
Other Study IDs: C22/18/008; S61997 (Other: Ethische commissie onderzoek UZ/KU Leuven)
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Healthy
Keywords: Healthy controls; Upper limb; Somatosensation; Sensory processing; Robotic assessment; Kinematics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Younger healthy adults: Healthy subjects in the age group of 18-30 years old, and without history of any neurological condition
- Older healthy adults: Healthy subjects aged 55 years and older, and without history of any neurological condition

SUMMARY:
After a stroke, more than two out of three patients experience problems with upper limb movement and sensation. During the past decade, robotic technology has been increasingly used to asses these problems in a detailed and accurate manner. However, sensory processing, one of the most important sensory functions, has not been assessed using robotic technology yet. Therefore, our group has developed a robotic assessment of sensory processing. This study is set up to obtain detailed information on how healthy controls perform on this task. This information can then help in identifying abnormal performances (i.e. upper limb sensory problems) in stroke patients. We aim to examine 40 healthy younger adults and 40 healthy older adults.

DETAILED DESCRIPTION:
Up to 70% of stroke survivors show upper limb impairments consisting of motor and/or somatosensory impairments. These impairments often persist well into the chronic stage, and may lead to significant limitations in activities of daily living and may negatively affect quality of life. It is therefore of utmost importance to accurately assess upper limb impairments. Clinical assessments exist for both motor and somatosensory function, but lack good psychometric properties. Robotic technology show promising potential and is readily available to assess motor function and proprioception. Robotic assessment for sensory processing is currently not yet available, despite being the most relevant somatosensory function. Indeed, sensory processing shows the strongest association with upper limb movement, and only shows incomplete recovery at 6 months after stroke.

Our group has recently developed a novel robotic assessment of sensory processing, using the Kinarm End-Point Lab (BKIN Technologies Ltd., Canada). This cross-sectional study is set up to collect a large amount of data from healthy controls, in order to obtain reference values for future research and to serve as control data for comparison with stroke patients. 40 younger healthy adults and 40 older healthy adults will be recruited and will undergo extensive clinical and robotic assessment of upper limb motor and somatosensory function, as well as cognitive function. This study also allows to investigate possible age-related decline in task performance, as well as investigation of the role of cognition in performance on this novel task.

ELIGIBILITY:
Inclusion Criteria:

- Aged 18-30 years old; or aged 55+

Exclusion Criteria:

* History of stroke or TIA
* Upper limb somatosensory and/or motor impairments
* Any serious musculoskeletal and/or other neurological conditions
* Serious communication or cognitive deficits
* No written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited from the community sample
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Kinarm: sensory processing task | Once in the chronic phase (at least 6 months after stroke)
  Newly-developed task on the Kinarm End-Point Lab used to assess passive and active sensory processing
Kinarm: working memory task | Once in the chronic phase (at least 6 months after stroke)
  Assessment of working memory on the Kinarm End-Point Lab, by asking the participant to remember the position of 3, 4, 5 or 6 targets simultaneously.

SECONDARY OUTCOMES:
Montreal cognitive assessment | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of cognitive function on an ordinal scale ranging from 0 to 30, with higher scores meaning better performance
Kinarm: position matching task | Once in the chronic phase (at least 6 months after stroke)
  Assessment of limb position sense using a 9-target mirror-matching task on the Kinarm End-Point Lab
Kinarm: visually guided reaching | Once in the chronic phase (at least 6 months after stroke)
  Assessment of motor function using a 4-target centre-out reaching task on the Kinarm End-Point Lab
Erasmus modified Nottingham sensory assessment | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of somatosensory function (including exteroception, proprioception and sensory processing) on an ordinal scale ranging from 0 to 40, with higher scores meaning better performance
Tactile discrimination test | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of sensory processing with an area under the curve based scoring system, with higher scores meaning better performance
Tactile functional object recognition | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of sensory processing on an ordinal scale ranging from 0 to 42, with higher scores meaning better performance
Stereognosis section of the original Nottingham sensory assessment | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of sensory processing on an ordinal scale ranging from 0 to 22, with higher scores meaning better performance
Wrist position sense test | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of wrist position sense on a continuous scale, with lower scores meaning better performance
Perceptual threshold of touch | Once in the chronic phase (at least 6 months after stroke)
  TENS-based assessment of exteroception on a continuous scale, with lower scores meaning better performance
Fugl-Meyer upper extremity assessment | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of motor function on an ordinal scale ranging from 0 to 66, with higher scores meaning better performance
Action research arm test | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of motor activity performance on an ordinal scale ranging from 0 to 57, with higher scores meaning better performance
Barthel index | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of activities of daily living on an ordinal scale ranging from 0 to 20, with higher scores meaning better performance
Star cancellation test | Once in the chronic phase (at least 6 months after stroke)
  Clinical assessment of visuospatial neglect on an ordinal scale ranging from 0 to 54, with higher scores meaning better performance, and a score below 44 indicating the presence of visuospatial neglect

CONTACTS AND LOCATIONS:
Overall Officials: Geert Verheyden, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided